CLINICAL TRIAL: NCT01225133
Title: The CARAKA-Trial: Complex Āyurvedic Treatment in Osteoarthritis of the Knee Against Standard Care.A Multicentre, Randomized, Controlled Clinical Trial Based on Traditional Āyurveda-Diagnosis.
Brief Title: Complex Āyurvedic Treatment in Osteoarthritis of the Knee Compared to Standard Care.
Acronym: CARAKA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Ministry of Health & Family Welfare, India (Other Government)
Responsible Party: Principal Investigator, Andreas Michalsen, Prof. Dr. med. Andreas Michalsen, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CARAKA-1
Record Dates: First submitted 2010-10-06; First posted 2010-10-20 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis, Osteoarthrosis, Arthritis, Arthrosis
MeSH Terms: conditions — Osteoarthritis; Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Complex Ayurvedic Treatment (Active Comparator): In the Āyurveda arm treatment will be individualized according to the Āyurveda diagnosis and include manual treatments, massages, dietary advice, specific consideration of selected food items, nutritional supplements, āyurvedic lifestyle and yoga posture advice and daily self-applied knee massage.
  Interventions: Other: Complex Ayurvedic Treatment; Other: Conventional Care
- Conventional Care (Active Comparator): Patients in the conventional standard care group will receive conventional standard care for OA of the Knee which includes self care advice, pain medication and intensified physiotherapy and follows the current international guidelines for OA of the knee.
  Interventions: Other: Complex Ayurvedic Treatment; Other: Conventional Care

INTERVENTIONS:
Other: Complex Ayurvedic Treatment — In the Āyurveda group treatment will be individualized according to the Āyurveda diagnosis and include manual treatments, massages, dietary advice, specific consideration of selected food items, nutritional supplements, āyurvedic lifestyle and yoga posture advice and daily self-applied knee massage.
Other: Conventional Care — Patients in the conventional standard care group will receive conventional standard care for OA of the Knee which includes self care advice, pain medication and intensified physiotherapy and follows the current international guidelines for OA of the knee.

SUMMARY:
The aim of this study is to evaluate the effectiveness of a complex āyurvedic diagnosis and treatment compared to conventional standard care in patients with OA of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients,
* Age 40-70 years,
* Prediagnosed, confirmed and documented diagnosis of OA of the knee. Diagnosis performed by a medical specialist (orthopedic surgeon, surgeon, radiologist) according to the American College of Rheumatology criteria,
* Documented radiologic changes of the knee-joint Kellgren-Lawrence criteria > or = grade 2 in conventional X-ray or MRI-scan,
* Mean average pain intensity of 40 or more on two 100 mm visual analogue scales in the 7 days before baseline assessment,
* Written informed consent.

Exclusion Criteria:

* Pain in the knee caused by oCongenital dysplasia of the affected knee oRheumatoid arthritis oAutoimmune diseases oMalignancies oStatus post Knee surgery oStatus post Arthroscopy
* Administration of chondroprotective drugs in the preceding 3 months,
* Intra-articular injection into the affected knee-joint during the preceding 3 months,
* Beginning of a systemic medication with corticosteroids within the preceding three months,
* Beginning of any new treatment for OA during the previous 4 weeks (with the exception of analgesic treatment with Paracetamol or NSAIDs),
* Pregnancy or breastfeeding,
* Acute mental disorders,
* Serious acute organic diseases,
* Serious chronic co-morbidity,
* Obesity WHO-grade II/III
* Blood coagulation disorders,
* Coagulation-inhibiting medication other than Aspirin and Clopidogrel,
* Invasive measures performed at the affected joint during the previous 12 weeks or planned within the following 12 month,
* In the process of applying for pension or disability benefits,
* Simultaneous participation in any other clinical trial,
* Participation in a clinical trial during the 6 month before inclusion into this trial,
* Missing of the written informed consent form.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-10; Primary Completion 2014-07 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster University Osteoarthritis Index (WOMAC) | week 12

SECONDARY OUTCOMES:
Western Ontario and McMaster University Osteoarthritis Index (WOMAC) Subscales | month 6
SF-36-questionnaire | week 12
POMS-questionnaire | week 12
Visual Analogue Scales: Pain | week 12
Visual Analogue Scales: Sleep | week 12
Western Ontario and McMaster University Osteoarthritis Index (WOMAC) Subscales | month 12
SF-36-questionnaire | month 6
SF-36-questionnaire | month 12
Western Ontario and McMaster University Osteoarthritis Index (WOMAC) Subscales | week 12
POMS-questionnaire | month 6
POMS-questionnaire | month 12

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof. Dr., Principal Investigator — Charité Medical University Berlin; Claudia M Witt, Prof. Dr., Principal Investigator — Charité University Medical Center Berlin
Locations (2):
- Germany (2):
  - Charité Medical University Cooperation Center Sonne und Mond, Berlin, State of Berlin
  - Immanuel Krankenhaus, Berlin, State of Berlin

REFERENCES:
- [Derived] Kessler CS, Dhiman KS, Kumar A, Ostermann T, Gupta S, Morandi A, Mittwede M, Stapelfeldt E, Spoo M, Icke K, Michalsen A, Witt CM. Effectiveness of an Ayurveda treatment approach in knee osteoarthritis - a randomized controlled trial. Osteoarthritis Cartilage. 2018 May;26(5):620-630. doi: 10.1016/j.joca.2018.01.022. Epub 2018 Feb 7. PMID 29426006
- [Derived] Witt CM, Michalsen A, Roll S, Morandi A, Gupta S, Rosenberg M, Kronpass L, Stapelfeldt E, Hissar S, Muller M, Kessler C. Comparative effectiveness of a complex Ayurvedic treatment and conventional standard care in osteoarthritis of the knee--study protocol for a randomized controlled trial. Trials. 2013 May 23;14:149. doi: 10.1186/1745-6215-14-149. PMID 23701973
- See also: Charite Medical University — http://www.charite.de